CLINICAL TRIAL: NCT00608777
Title: Effect of Topical Calcipotriene/Betamethasone (Taclonex) in Managing Localized Mild Breakthrough in Moderate to Severe Plaque Psoriasis Patients Receiving Efalizumab ( Raptiva).
Brief Title: Effect of Topical Calcipotriene/Betamethasone (Taclonex) in Managing Localized Breakthrough in Moderate to Severe Plaque Psoriasis in Patients Receiving Efalizumab (Raptiva)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawal of marketing autorization of efalizumab by the EMEA.
Sponsor: Derm Research, PLLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Leon Kircik, M.D., Principal Investigator, Derm Research, PLLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACD4311s
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Plaque Psoriasis
Keywords: Localized mild breakthrough
MeSH Terms: interventions — calcipotriene; Betamethasone; betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Calcipotriene/betamethasone — One application to affected areas, once a day for two weeks. The PI may choose to extend treatment until Week 4 if necessary.
  Other Names: Taclonex

SUMMARY:
The purpose of this study is to determine if calcipotriene/bethamethasone can safely and effectively manage the occurence of LMB (mild localized breakthrough) in patients recieving efalizumab (Raptiva) for moderate to severe plaque psoriasis.

It is hypothesized that calcipotriene/betamethasone (Taclonex) could be used to manage LMB and thus allow patients to continue efalizumab without interruption.

DETAILED DESCRIPTION:
LMB (localized mild breakthrough)is one of two psoriasis adverse events commonly seen in efalizumab treated patients. It is generally papular in nature and does not involve existing lesions. Clinical experience suggests that LMB may not have a clinical impact in patients responding to efalizumab and therefore may be treated without interrupting efalizumab therapy. To relieve discomfort topical therapy may be indicated until the symptoms are resolved.

This is a single arm, open label study. Fifteen patients who are receiving efalizumab before entrance into this study and who develop LMB wil be enrolled. Topical calcipotriene/betamethasone (Taclonex) will be applied to the areas (except face, axillae or groin) once a day for two weeks. The PI may choose to continue two more weeks if needed for a total of four weeks of therapy. All patients will continue with efalizumab without dose modification for the duration of the study. Patients will return for follow up visits at weeks 2, 4 and 6. Topical desonide may be used for LMB involvement of the face, groin or axillae.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written, informed consent and comply with study assessments for the full duration of the study.
* Age 18 years or older.
* Moderate to severe plaque psoriasis being treated with efalizumab.
* Develop LMB during efalizumab treatment.
* PGA of LMB at least mild (2) excluding face, axillae and groin.

Exclusion Criteria:

* Patients with known hypersensitivity to efalizumab, calcipotriene/betamethasone or any of its components.
* Pregnant or lactating women.
* Known or suspected disorders of calcium metabolism.
* Erythrodermic, exfoliative and/or pustular psoriasis.
* Concomitant use of topical thaerapy, phototherapy or immunosuppressive agents.
* LMB (in areas other than face, axillae or groin) constitutes more than 30% of total body surface area.
* Patients with generalized inflammatory flare which is defined as widespread worsening of psoriasis characterized by erythematous and and edematous lesions within exisiting plaques.
* Any other condition the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H Kircik, M.D., Principal Investigator — DermResearch, PLLC
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

REFERENCES:
- [Background] de Jong EM. The course of psoriasis. Clin Dermatol. 1997 Sep-Oct;15(5):687-92. doi: 10.1016/s0738-081x(97)00023-0. No abstract available. PMID 9313967
- [Background] Carey W, Glazer S, Gottlieb AB, Lebwohl M, Leonardi C, Menter A, Papp K, Rundle AC, Toth D. Relapse, rebound, and psoriasis adverse events: an advisory group report. J Am Acad Dermatol. 2006 Apr;54(4 Suppl 1):S171-81. doi: 10.1016/j.jaad.2005.10.029. PMID 16488339
- [Background] Menter A, Leonardi CL, Sterry W, Bos JD, Papp KA. Long-term management of plaque psoriasis with continuous efalizumab therapy. J Am Acad Dermatol. 2006 Apr;54(4 Suppl 1):S182-8. doi: 10.1016/j.jaad.2005.10.028. No abstract available. PMID 16488340
- [Background] Werther WA, Gonzalez TN, O'Connor SJ, McCabe S, Chan B, Hotaling T, Champe M, Fox JA, Jardieu PM, Berman PW, Presta LG. Humanization of an anti-lymphocyte function-associated antigen (LFA)-1 monoclonal antibody and reengineering of the humanized antibody for binding to rhesus LFA-1. J Immunol. 1996 Dec 1;157(11):4986-95. PMID 8943405
- [Background] Raptiva Prescribing Information. Genentech, Inc. June 2005
- [Background] Taclonex Prescribing Information. Warner Chilcott (US), Inc. Jan 2006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from January 2008 through December 2008. Subjects recruited from physician data base.
Pre-assignment Details: Subjects experiencing mild localized breakthrough associated with Raptiva use were recruited.
Period: Overall Study
Arm/Group | Open Label Taclonex
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Taclonex
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Acheive a Score of Clear (0) or Almost Clear (1) on the PGA of LMB at Week 2
Time Frame: week 2
Arm/Group | Open Label Taclonex
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Open Label
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Study terminated due to withdrawal of Raptiva from the market. Study specifically designed to address a side effect associated with the administration of Raptiva. Therefore no data analysis completed for this study and no measuremnet of outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes